CLINICAL TRIAL: NCT03246997
Title: Project Powerfood: Promoting Food Security, Equity, and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: New York Common Pantry (Unknown); Corbin Hill Food Project (Unknown); Wholesome Wave (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 16-0031
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Obesity
Keywords: Food Insecure
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Intervention Model Description: Participants are enrolled in the study and randomly assigned to the immediate intervention or the delayed intervention group. Participants in the immediate intervention group will receive the intervention for 6 months with a 6-month and 12-month follow-up starting from day one of enrollment. Participants in the delayed intervention group will receive the intervention beginning 6 months after enrollment with a 6-month and 12-month follow-up starting from day one of enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autumn Group (Other): Intervention Group
  Interventions: Other: Autumn Group
- Spring Group (Other): Delayed Intervention
  Interventions: Other: Spring Group

INTERVENTIONS:
Other: Autumn Group — The intervention is participating in a fruit and vegetable farm share for 6 months.
  Other Names: Fresh fruit and vegetable subsidy
  Arms: Autumn Group
Other: Spring Group — The intervention is participating in a fruit and vegetable farm share for 6 months.
  Other Names: Fresh fruit and vegetable subsidy
  Arms: Spring Group

SUMMARY:
Project Powerfood is a pilot program aimed at addressing food insecurity and food access in primary care through the implementation of a food prescription program in collaboration with a number of community partners. The objectives of this project are:

1. Implement screening for food insecurity in adult and pediatric primary care practices at Mount Sinai.
2. Provide fresh fruit and vegetable "prescriptions" to be redeemed for farm shares from local partner, the Corbin Hill Food Project. Prescriptions will provide 50% off of a fruit and vegetable box. Participants will have the option to purchase 2 boxes per month for 6 months.
3. Pilot prescriptions with 50 adult patients with poorly-controlled diabetes and 50 obese children who are food insecure and/or receive SNAP and/or WIC benefits. Examine/evaluate:

   1. Feasibility of program in a busy primary care practice
   2. Outcomes before and after the intervention (at baseline, 6 and 12 months), including diet, diabetes control, and body mass index (BMI)
   3. Outcomes in a comparison group (that will receive the food prescriptions beginning at 6 months)

ELIGIBILITY:
Inclusion Criteria:

* Food insecure and/or receive SNAP and/or WIC
* Adult patients: poorly-controlled diabetes (hemoglobin A1c greater than 8.0%)
* Pediatric patients: obesity, ages 5-11
* Speak English or Spanish

Exclusion Criteria:

* Food secure and do not receive SNAP or WIC
* Adult Patients: do not have diabetes
* Pediatric Patients: not obese, under 5 years old or between 11 and 18
* Speak neither English or Spanish
* Severe kidney disease (Chronic Kidney Disease (CKD Stage IV or V)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Number of farm shares picked-up | up to 12 months
  Number of farm shares picked-up
Overall satisfaction score | up to 12 months
  overall satisfaction with the program measured by likelihood of recommending the program to a friend on a 4 point scale 1 = not likely at all, 2 = somewhat likely, 3 = likely 4 = very likely

SECONDARY OUTCOMES:
Health Eating Index | up to 12 months
  Diet quality, defined by the Health Eating Index which will be derived from the completion of 2 24-hour dietary recalls
BMI | up to 12 months
  The child participant's body mass index
USDA US Household Food Security Survey | up to 12 months
  Food Insecurity as measured by an 18-item Self reported concern about being able to afford food or have access to food at the end of a given month. Responses to the questions in the food security survey module are combined into a scale using non-linear statistical methods based on the Rasch measurement model.
Hemoglobin A1c level | up to 12 months
  The adult participant's glycemic control (as measured by hemoglobin A1c)
The Stanford Patient Education Research Center Diabetes Self-Efficacy Scale | up to 12 months
  Diabetes Self Efficacy as measured by Self reported feelings on one's ability to control and manage their diabetes. 8-item survey, total range from 8 (not at all confident) to 80 (totally confident).
Self Efficacy for Eating/Cooking Fruit and Vegetables by Condrasky | up to 12 months
  Cooking attitudes as measured by self reported attitudes about cooking and the use of the provided fresh fruits and vegetables to provide food to themselves and or their families.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Mayer, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No